CLINICAL TRIAL: NCT06392308
Title: The Impact of Smoking on Postoperative Delirium and Recovery Quality in Elderly Surgical Patients
Brief Title: The Impact of Smoking on the Prognosis of Elderly Surgical Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Chaochao Zhong, Principal Investigator, Affiliated Hospital of Nantong University
Other Study IDs: 2023-K213-01
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Delirium, Postoperative
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoker group: who smoke more than one cigarette per day continuously or cumulatively for six months; more than four times a week but averaging less than one cigarette per day
  Interventions: Other: none intervention
- Non-smoker group: never smoke
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention — No interventions are administered to either group of patients.

SUMMARY:
Postoperative delirium is a common complication that frequently occurs in elderly patients after surgery. It not only increases the length of hospital stays and healthcare costs but also raises the incidence of postoperative cognitive dysfunction and even mortality. However, the underlying mechanisms of its onset are not yet fully understood. Evidence suggests that smoking can lead to gut microbiota dysbiosis and metabolic dysfunction, and the gut microbiota and its metabolites play a crucial role in cognitive function through the gut-brain axis. Yet, no studies have reported whether smoking could affect the occurrence of postoperative delirium and the quality of postoperative recovery through the gut microbiota. This study aims to observe the incidence of postoperative delirium and the postoperative recovery quality scores between smokers and non-smokers.

DETAILED DESCRIPTION:
After obtaining approval from the ethics committee, patients are recruited, informed of the trial process and potential risks, and their informed consent is obtained and signed. According to the WHO definition, patients are classified into smokers (defined as those who smoke more than one cigarette per day continuously or cumulatively for six months; more than four times a week but averaging less than one cigarette per day) and non-smokers (never smoked). Fecal and blood samples are collected from both groups of patients preoperatively, and perioperative data is gathered. Postoperatively, an uninformed observer assesses the patients for delirium and recovery quality.

ELIGIBILITY:
Inclusion Criteria:

* Age >60 years;
* American Society of Anesthesiologists (ASA) preoperative anesthesia classification ASA Grades I and II;
* Undergoing elective surgery;
* Patients and their families are able to understand and complete various scoring scales and voluntarily sign informed consent.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score <23;
* Preoperative biochemical tests indicate renal dysfunction or active liver disease;
* History of definite neurological or psychiatric disorders or history of taking corresponding medications before surgery;
* History of alcohol abuse or drug dependency;
* Taking antidepressant medications;
* American Society of Anesthesiologists (ASA) preoperative anesthesia classification > Grade II.

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elderly patients who meet the inclusion criteria are divided into a smoking group and a non-smoking group based on their smoking status. The general information of the patients, perioperative data, and postoperative follow-up data are recorded. By conducting propensity score matching analysis, differences in outcomes due to confounding factors are minimized, and exploratory analysis is performed on the matched patient data to investigate the impact of gut microbiota and metabolism on the incidence of postoperative delirium and the quality of postoperative recovery.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | Within 3 days post-surgery
  CAM method
Quality of recovery in the first postoperative day | Up to 24 hours after surgery.
  Quality of recovery is assessed with the Quality of Recovery-15 questionaire in the first postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chao Zhong, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No